CLINICAL TRIAL: NCT05955937
Title: ImpleMEntation of a Digital-first Care deLiverY Model for Heart Failure in Uganda
Acronym: MEDLY Uganda
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000035428; R01HL166585 (NIH)
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: After 1-2 month-long run-in periods to allow for integration and adoption of the interventions all sites will receive the multi-component implementation strategy, beginning with the Core HF and followed by Medly Uganda. Sites will be randomized using a randomization software to receive the interventions at different start points after the first six months, for varying durations throughout the 3-year study period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Step 1. Core HF intervention period (Experimental): All sites will be trained in an evidence-based clinical care bundle for HF, to ensure standardized basic HF care across the participating RRHs in the study. For this service bundle which will augment self-care (Core-HF), the investigators will train providers in an evidence-based HF clinical care service bundle including a care protocol (treatment algorithm for HF), self-care training for patients and providers, and medication stock management prior to introducing the digital health intervention (Medly Uganda, described in Arm 2).
  Interventions: Other: Enhanced HF Clinical Care (Core-HF)
- Step 2. Core-HF plus Medly Uganda digital health intervention (Experimental): Medly Uganda will utilize a patient-facing mobile health application designed to improve self-care among patients with HF. Its principal components are: 1) a patient-facing mobile application that processes patient-reported symptoms and generates algorithm-driven messages to guide self-care and symptom management and 2) a clinician- facing internet dashboard that monitors symptom reports and facilitates nurse-guided management recommendations and physician backup support. The project will support an integrated, digital interface at participating hospitals to monitor and intervene with patients who are using the mobile health application.
  Interventions: Other: Digital health intervention (Medly Uganda) plus enhanced HF clinical care (Core-HF)

INTERVENTIONS:
Other: Enhanced HF Clinical Care (Core-HF) — All clinical care providers involved in HF care at participating RRHs will be trained in a HF service bundle including a care protocol (treatment algorithm based on global guidelines), self-care training for patients and providers, and medication stock management to ensure supply of HF medications to patients in need.
  Arms: Step 1. Core HF intervention period
Other: Digital health intervention (Medly Uganda) plus enhanced HF clinical care (Core-HF) — A patient-facing mobile health application designed to improve self-care will be provided to the study participant, which will operate on all mobile devices. This will be introduced after the Core-HF intervention has been delivered.
  Arms: Step 2. Core-HF plus Medly Uganda digital health intervention

SUMMARY:
This is a stepped wedge, cluster-randomized study, that will implement a digital-first, multi-component strategy for Heart Failure (HF) to improve HF self-care at 6 Regional Referral Hospital (RRH) outpatient departments in Uganda. The investigators will evaluate both implementation and clinical outcomes using mixed methods. . First, investigators will assess the implementation and clinical effectiveness of an enhanced standard-of-care clinical bundle, and a digital health intervention to improve HF self-care in Uganda (Aim 1). To do this, the investigators will conduct a stepped-wedge, cluster randomized trial that includes a brief control period followed by a clinical care service bundle for HF (Core HF), followed by the introduction of the digital health application (Medly Uganda). The co-primary outcomes will be the Self-Care of HF Index (implementation) and the composite of mortality and HF hospitalization (clinical effectiveness).

To ensure standardized basic HF care which will augment self-care, investigators will train providers in an evidence-based HF clinical care service bundle (Core HF) including a care protocol (treatment algorithm for HF), self-care training for patients and providers, and medication stock management prior to the introduction of the digital health intervention (Medly Uganda). Medly Uganda will utilize a patient-facing mobile health application designed to improve self-care among patients with HF. Its principal components are: 1) a patient-facing mobile application that processes patient-reported symptoms and generates algorithm-driven messages to guide self-care and symptom management and 2) a clinician-facing internet dashboard that monitors symptom reports and facilitates nurse-guided management recommendations and physician backup support. The project supports an integrated, digital interface at participating hospitals to monitor and intervene with patients using the mobile health application.

DETAILED DESCRIPTION:
In parallel to the above, the investigators will conduct a mixed methods process evaluation to inform iterative adjustments to the implementation processes, i.e., a Learn- As-You-Go design by reviewing qualitative feedback and quantitative intervention data (Aim 2). Then, cost effectiveness, and sustainability factors for Medly Uganda, including an examination of cost, cost-effectiveness, and equity of Medly Uganda from a financial and societal perspective will be explored (Aim 3).

The focus of this registration will be Aim 1 and Aim 2.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of New York Heart Association (NYHA) Class II-III HF
* Access to a mobile phone
* Basic reading skills in 1 of the offered languages, as determined by their clinical care provider. Languages will include: Lugbara in Arua, Lugiso in Mbale, Runyankole in Mbarara, Luganda in Masaka, Rutooro in Fort Portal, and Langi in Lira in addition to English.

Exclusion Criteria:

* Any individual not meeting the above inclusion criteria
* Inability to provide informed consent, as determined by the nurse manager
* Active medical condition requiring hospitalization, such as cardiac ischemia (acute electrocardiographic changes and/or positive biomarkers, if available), syncope, or significant fluid overload
* Echocardiography findings that do not support a diagnosis of HF as determined during a study visit. This exclusion might occur following enrollment and new patients may be consented and enrolled to compensate for these exclusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change in Self-Care of Heart Failure Index (SCHFI) | baseline, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  The SCHFI v7.23 is a validated 39-item instrument hat assesses maintenance, management, and self-confidence of heart failure self-care. Scores range from 0-100 with higher scores indicating improved self care.
Clinical Effectiveness | baseline, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  A composite of the number of participants with mortality and HF hospitalization will be used to assess clinical effectiveness. This outcome is the most widely used composite clinical endpoint in HF trials globally.

SECONDARY OUTCOMES:
Participant fidelity to self-care assessed by medication adherence using Medication Adherence Report Scale (MARS-5) and 7-day recall | up to 36 months
  Participant fidelity will be assessed by self report administered by the Research Assistant. The MARS-5 is a 5-item questionnaire that asks the frequency of behaviors that indicate non-adherence (forgetting to take medications, for example). The range of score is 5-25. A higher score indicates higher adherence (positive outcome of self-care).
Change in NYHF Classification | up to 36 months
  As assessed by clinical care provider, heart failure as measured by the New York Heart Failure Classification 1. Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc. 2. Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity. 3. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances. Comfortable only at rest, and 4.Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients. Lower classes indicate a positive outcome.
Change in 6-minute walk test | baseline, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  The 6-minute walk test monitors physical conditioning. It measures the distance an individual can walk over a total of six minutes on a hard, flat surface. The individual can self-pace and rest as needed as they walk back and forth along a marked course. The participant can use an assistive walking device they normally use, such as a cane. The minimum clinically important difference in 6-minute walk distance is approximately 30 meters, a difference that is associated with mortality.
Change in Pro-NT Brain Natriuretic Peptide (Pro-NT BNP) | baseline, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  Levels of Pro-NT BNP, a widely used prognostic marker in HF, will be measured in blood samples in pg/mL. Lower values indicate a positive outcome.
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) | baseline, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  The KCCQ is a 12-item questionnaire that measures symptoms, physical and social limitations, and quality of life in participants with heart failure. KCCQ scores are scaled from 0 to 100, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
Change in EuroQol -5D (EQ-5D) | baseline, 6 months, 12 months, 18 months, 24 months, 30 months and 36 months
  EQ-5D 5L is a standardized participant completed questionnaire that measures health-related quality of life. It is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3=moderate problems, 4= severe problems, and 5= extreme problems. Higher scores indicated greater levels of problems across each of the five dimensions. A utility score was obtained by using a weighted combination of the levels of the five dimension-scales.
Facility fidelity to implementation strategy assessed by vital sign checks and other intervention components | up to 36 months
  Percentage of patients receiving Core HF components (i.e., vital sign checks; self-care guidance) based on the penultimate implementation strategy
Facility fidelity to implementation strategy assessed by the availability of medications | up to 36 months
  Facility fidelity to implementation strategy will be assessed by the prescribing-to-dispensing ratio of HF medications at facility pharmacy

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Schwartz, MD, Principal Investigator — Yale University; Isaac Ssinabulya, MD, Principal Investigator — Uganda Initiative for Integrated Management of Non-Communicable Diseases (UINCD); Joseph Cafazzo, PhD, Principal Investigator — University Health Network of Toronto
Locations (7):
- Uganda (7):
  - Arua Regional Referral Hospital, Arua
  - Fort Portal Regional Referral Hospital, Fort Portal
  - Uganda Heart Institute, Kampala
  - Lira Regional Referral Hospital, Lira
  - Masaka Regional Referral Hospital, Masaka
  - Mbale Regional Referral Hospital, Mbale
  - Mbarara Regional Referral Hospital, Mbarara

IPD SHARING:
Plan to Share IPD: No